CLINICAL TRIAL: NCT05591690
Title: Use of MiniMed 780G System in Children and Adolescents, a French Real Life Observational Study
Brief Title: Use of MiniMed 780G System in Children and Adolescents
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL22_0420
Record Dates: First submitted 2022-09-21; First posted 2022-10-24 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Diabetes
Keywords: Advanced hybrid closed loop; pediatrics; real-world; time in range
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hybrid closed-loop technology have shown that it improves glycemic control parameters, but the investigators do not have sufficient data at more than 6 months of follow-up, allowing us to describe the effectiveness of these systems in the long term.

All MiniMed 780G system users from November 2020 to March 2022 were included (n=32) For every time points, there was a significant difference in Time In Range between the pre-AHCL and post-AHCL. Noted difference were +14.5% and, +10.8% at respectively 3 months and 1 year. No more hypoglycemia were identified.

This "real-life" analysis shows that the algorithm is effective in improvement of metabolic control for T1 diabetic children and adolescents, at one year of follow-up.

However, an effect of breathlessness is observed which underlined the need for a solid therapeutic education program.

ELIGIBILITY:
Inclusion criteria:

All children with type 1 diabetes in whom a Medtronic G780 closed-loop pump was placed between November 2020 and March 2022 in our center were included.

Exclusion criteria:

Participant opposition

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Diabetic minors treated with closed-loop insulin pumps
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Glycated hemoglobin | 1 year
  Percentage of glycated hemoglobin measured by the MiniMed 780G system
Time spent in range Level with glucose levels within the norm | 1 year
  Time spent with glucose levels between 70 and 180 mg/dL
Time spent with glucose levels below range | 1 year
  Time spent with glucose levels inferior to 70mg/dL
Time spent with glucose levels above range | 1 year
  Time spent with glucose levels superior to 180 mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Fabienne Dalla Vale, PH, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC